CLINICAL TRIAL: NCT00626626
Title: Clofarabine and Non-Myeloablative Allogeneic Hematopoietic Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, David F. Claxton, MD, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25223
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-03

CONDITIONS: Leukemia; Myelodysplastic Syndrome; Chronic Myelogenous Leukemia; Lymphoma; Hodgkin's Lymphoma; Multiple Myeloma
Keywords: leukemia; myelodysplastic syndrome; chronic myelogenous leukemia; lymphoma; mantle cell lymphoma
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma; Hodgkin Disease; Multiple Myeloma; Lymphoma, Mantle-Cell | interventions — sodium tetrametaphosphate; Alemtuzumab; Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- "Clofar, Cyclophos, Alemtuzumab" (Experimental): Phase 1: 1-3 patients will be treated in order to establish Cyclophosphamide and Clofarabine dose and to confirm reasonable safety and engraftment efficacy.
  Drug - Clofarabine,Cyclophosphamide & Alemtuzumab - Clofar (30mg/m2) D -8 to -4; Cyclo (500mg/m2) D -8 & -7 & Alem (20mg over 2hrs)
  Interventions: Drug: Clofar, Cyclophos, Alemtuzumab
- "Clofar, Cyclophos,Alemtuzumab(Ph II)" (Experimental): Phase II patients 4-9 will treat at the selected dose level of Clofarabine and Cyclophosphamide.
  Drug - Clofarabine, Cyclophosphamide & Alemtuzumab Clofar (30mg/m2) D -8 to -4; Cyclo (1000mg/m2) D -8 & -7 & Alem (20mg)-pts.
  Interventions: Drug: Clofar, Cyclophos,Alemtuzumab(Ph II)

INTERVENTIONS:
Drug: Clofar, Cyclophos, Alemtuzumab — Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 500 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion.
  Other Names: CLOLAR
  Arms: "Clofar, Cyclophos, Alemtuzumab"
Drug: Clofar, Cyclophos,Alemtuzumab(Ph II) — Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 1000 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion (patients 4-9)
  Other Names: Clolar; Campath
  Arms: "Clofar, Cyclophos,Alemtuzumab(Ph II)"

SUMMARY:
Allogeneic hematopoietic transplant is curative for many patients with hematological neoplasms but conditions to provide optimal engraftment and anti-tumor efficacy with minimal toxicity are still under way. Clofarabine is a newly licensed agent with dramatic anti-leukemic activity. Its incorporation into a regimen for pre-transplant conditioning of acute leukemia and lymphoma patients is logical, exploiting both the anti-tumor activities it is recognized to have and the immunosuppressive activity seen with drugs in its class.

DETAILED DESCRIPTION:
Non-myeloablative conditioning allows curative allogeneic hematopoietic transplantation for patients unable to tolerate more toxic conventional conditioning regiments. These regiments continue to be refined and evolve. No standard regimen is yet agreed upon. The incorporation of the newly licenses agent Clofarabine into a non-myeloablative regimen is logical given its recognized anti-leukemic activity. This study will assess the safety and efficacy of Cyclophosphamide and Clofarabine in promoting hematopoietic engraftment after allogeneic transplant of blood stem cells. Patients eligibility will include those with advanced hematological neoplasms who might benefit from allogeneic blood cell transplant. Patients must have adequate organ function and suitable related or unrelated donors for transplant. In Phase I of the study 9-12 patients will be treated in order to establish Cyclophosphamide and Clofarabine dose, and to confirm reasonable safety and engraftment efficacy. Phase II will treat at total of 20 patients at the selected dose level of Clofarabine and Cyclophosphamide. Results will be compared to extensive Penn State Milton S. Hershey Medical Center experience using Fludarabine and Cyclophosphamide in a similar patient population. Supportive care, including graft versus host disease prophylaxis will be similar to that recently used at Hershey Medical Center. Primary endpoints will include survival and engraftment as compared to historical results at Hershey Medical Center. Disease specific outcomes for frequent diagnoses such as acute leukemia and non-hodgkin's lymphoma will be assessed as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

Phase I

* Acute leukemia - secondary or beyond first remission or in CR with poor risk cytogenetics, myelodysplastic syndrome IPPS Int-2 or high risk, chronic myelogenous leukemia in accelerated or blast crisis and imatinib refractory or lymphoma having failed second line therapy or relapsed mantle cell lymphoma.

Phase II

* Acute leukemia secondary or at high risk for relapse, myelodysplastic syndrome IPPS Int-2 or high risk or having failed other therapy, chronic myelogenous leukemia, lymphoma having failed first line therapy or at high risk, relapsed Hodgkin's, CCL progressed beyond initial therapy, multiple myeloma beyond initial response or with high risk features.
* Must have an HLA matched or 5/6 matched related donor at at least a 5/6 matched unrelated donor available.
* Have adequate renal and hepatic functions
* Capable of understanding the investigational nature, potential risk and benefits of the study and able to provide valid informed consent.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients of childbearing potential must use an effective contraceptive method during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy or immunotherapy other than as specified in the protocol.
* Use of investigational agents within 30 days and no cytotoxic anticancer agents within 2 weeks before study entry with the exception of hydroxyurea. The patient must have recovered from all non-hematological acute toxicities from any previous therapy.
* Other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo treatment.
* Patients with systemic fungal, bacterial, viral, or other infection not controlled.
* Pregnant or lactating patients.
* Any significant concurrent disease, illness or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow-up or interpretation of study results.
* Age > 70 (for Phase 1) or 75 (for Phase 2)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David F Claxton, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karch J, Zhu J, Ehmann WC, Claxton D. Clofarabine and CY do not yield reliable engraftment of hematopoietic stem cells. Bone Marrow Transplant. 2012 Aug;47(8):1134-5. doi: 10.1038/bmt.2011.224. Epub 2011 Nov 14. No abstract available. PMID 22080968

RESULTS

PARTICIPANT FLOW:
Groups:
- "Clofar, Cyclophos, Alemtuzumab": Phase 1: 1-3 patients will be treated in order to establish Cyclophosphamide and Clofarabine dose and to confirm reasonable safety and engraftment efficacy.
  Dose Level I: Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 500 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion.
- "Clofar, Cyclophos,Alemtuzumab(Ph II)": Phase II patients 4-9 will treat at the selected dose level of Clofarabine and Cyclophosphamide.
  Dose Level 2: Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 1000 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion (patients 4-9)
Period: Overall Study
Arm/Group | "Clofar, Cyclophos, Alemtuzumab" | "Clofar, Cyclophos,Alemtuzumab(Ph II)"
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level1: Phase 1: 1-3 patients will be treated in order to establish Cyclophosphamide and Clofarabine dose and to confirm reasonable safety and engraftment efficacy.
  Dose Level I: Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 500 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion.
- Dose Level 2: Phase II patients 4-9 will treat at the selected dose level of Clofarabine and Cyclophosphamide.
  Dose Level 2: Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 1000 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion (patients 4-9)
- Total: Total of all reporting groups
Arm/Group | Dose Level1 | Dose Level 2 | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Engraftment of Allogeneic Blood Cells.
Description: Establish the safety of Clofarabine and cyclophosphamide preceding allogeneic hematopoietic engraftment. Assess the efficacy of Clofarabine and cyclophosphamide as conditioning for promoting allogeneic hematopoietic engraftment.
  Adequacy of engraftment will be assessed via assessment of chimerism (percent donor engraftment). Less than 20% engraftment by day 30 is then failure of engraftment.
  Safety is defined per common toxicity criteria - Non-Hematological and non renal toxicities of ≥grade 3 or ≥grade 4 up to day 30 are scored as toxicity.
Time Frame: two years
Measure: Count of Participants; unit: Participants
Groups:
- Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I ): Phase 1: 1-3 patients will be treated in order to establish Cyclophosphamide and Clofarabine dose and to confirm reasonable safety and engraftment efficacy.
  Dose Level I: Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 500 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion.
- Clofarabine, Cyclophosphamide & Alemtuzumab (Phase II): Phase II patients 4-9 will treat at the selected dose level of Clofarabine and Cyclophosphamide.
  Dose Level 2: Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 1000 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion (patients 4-9)
Arm/Group | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I ) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase II)
Number analyzed (Participants) | 5 | 3
Participants
  Adequate Engraftment | 2 | 1
  Safety | 5 | 3

2. Secondary Outcome: Disease-Free Survival
Description: Observe disease free survivals in acute leukemia and lymphoma patients receiving allogeneic hematopoietic transplant after Clofarabine and cyclophosphamide conditioning.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Groups:
- Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I): Phase 1: 1-3 patients will be treated in order to establish Cyclophosphamide and Clofarabine dose and to confirm reasonable safety and engraftment efficacy.
  Dose Level I: Hydrocortisone 100 mg IV 30 minutes prior to each dose of Clofarabine. Ondansetron 16 mg PO or IV or another comparable antiemetic should be given prior to each dose of Clofarabine. An additional similar dose should be given prior to Cyclophosphamide dose. Clofarabine 30 mg/M2 -8 through - 4 (5 doses) infusion. Alemtuzumab on day -8 only and after Clofarabine. Cyclophosphamide 500 mg/m2 Days -8 and -7 (2 doses) given over 1 hour beginning 4 hours after the beginning of Clofarabine infusion.
Arm/Group | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase II)
Number analyzed (Participants) | 5 | 3
Participants
  Disease Free | 0 | 1
  Relapsed | 5 | 2

3. Secondary Outcome: Overall Survival
Description: Observe overall survival in leukemia and lymphoma patients receiving transplant after clofarabine and cyclophosphamide conditioning.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I ) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase II)
Number analyzed (Participants) | 5 | 3
Participants
  Survival (2 years) | 1 | 1
  Lost to Followup | 1 | 0
  Died | 3 | 2

ADVERSE EVENTS:
Arm/Group | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase II)
Serious Adverse Events (participants affected / at risk) | 4/5 | 1/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I) (N=5) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase II) (N=3)
Failure to engraft (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase I) (N=5) | Clofarabine, Cyclophosphamide & Alemtuzumab (Phase II) (N=3)
Decreased Leukocytes (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Decreased ANC (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 5 (7) | 3 (4)
Decreased Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Skin (due to shingles) (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (6) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 2 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less